CLINICAL TRIAL: NCT02527798
Title: Safety of Furosemide in Premature Infants at Risk of Bronchopulmonary Dysplasia
Brief Title: Safety of Furosemide in Premature Infants at Risk of Bronchopulmonary Dysplasia (BPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Duke University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 15-1978; HHSN27500033 (Other Grant/Funding Number: National Institute of Child Health and Human Development (NICHD)); HHSN27500035 (Other Grant/Funding Number: NICHD); 5R01FD005101-02 (FDA)
Record Dates: First submitted 2015-08-04; First posted 2015-08-19 (Estimated); Results first posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-09

CONDITIONS: Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Furosemide Cohort 1 (Experimental): Within cohort 1, infants will be randomized using a 3:1 scheme to receive furosemide or placebo. Those randomized to receive furosemide will receive (1mg/kg daily intravenously or 2 mg/kg daily enterally for 28 days.
  Interventions: Drug: Furosemide Cohort 1
- Placebo Cohort 1 (Placebo Comparator): Infants randomized to the placebo treatment group will receive the equivalent volume of dextrose 5% for IV use or enteral use (if receiving enteral study drug).
  Interventions: Other: Placebo
- Furosemide Cohort 2 (Experimental): Cohort 2 Infants will receive furosemide (1mg/kg every 6 hours intravenously or 2 mg/kg every 6 hours daily enterally) for 28 days.
  Interventions: Drug: Furosemide Cohort 2
- Furosemide Cohort 3 (Experimental): Cohort 3 Infants will receive furosemide (2mg/kg every 6 hours intravenously or 4 mg/kg every 6 hours daily enterally) for 28 days.
  Interventions: Drug: Furosemide Cohort 3
- Placebo Cohort 2 (Placebo Comparator): Infants randomized to the placebo treatment group will receive the equivalent volume of dextrose 5% for IV use or enteral use (if receiving enteral study drug).
  Interventions: Other: Placebo
- Placebo Cohort 3 (Placebo Comparator): Infants randomized to the placebo treatment group will receive the equivalent volume of dextrose 5% for IV use or enteral use (if receiving enteral study drug).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Furosemide Cohort 1 — furosemide 1 mg/kg q 24 hours IV or 2 mg/kg q 24 hours enterally Cohorts will be enrolled sequentially after a safety review.
  Other Names: Lasix
  Arms: Furosemide Cohort 1
Drug: Furosemide Cohort 2 — furosemide 1 mg/kg q 6 hours IV or 2 mg/kg q 6 hours enterally Cohorts will be enrolled sequentially after a safety review.
  Other Names: Lasix
  Arms: Furosemide Cohort 2
Drug: Furosemide Cohort 3 — furosemide 2 mg/kg q 6 hours IV or 4 mg/kg q 6 hours enterally Cohorts will be enrolled sequentially after a safety review.
  Other Names: Lasix
  Arms: Furosemide Cohort 3
Other: Placebo — Sugar water will be administered in a equivalent volume as drug intervention.
  Other Names: sugar water
  Arms: Placebo Cohort 1; Placebo Cohort 2; Placebo Cohort 3

SUMMARY:
This study will describe the safety of furosemide in premature infants at risk of bronchopulmonary dysplasia and determine the preliminary effectiveness and pharmacokinetics (PK) of furosemide. Funding Source - FDA OOPD

DETAILED DESCRIPTION:
Infants will receive a placebo or furosemide for 28 days. Blood samples will be collected for pharmacokinetic analysis.Premature infants will be randomized to receive placebo or furosemide in a dose escalating approach.

Follow up information will be collected up to 7 days after the last dose and at 36 weeks post menstrual age. The final study assessment will occur at the time of discharge, early termination or transfer.

ELIGIBILITY:
Inclusion Criteria:

1. Receiving positive airway pressure (nasal continuous airway pressure, nasal intermittent positive pressure ventilation, or nasal cannula flow > 1LPM) or mechanical ventilation (high frequency or conventional)
2. < 29 weeks gestational age at birth
3. 7-28 days postnatal age at time of first study dose

Exclusion Criteria:

1. Exposure to any diuretic ≤ 72 hours prior to first study dose
2. Previous enrollment and dosing in current study, "Safety of Furosemide in Premature Infants at Risk of Bronchopulmonary Dysplasia"
3. Hemodynamically significant patent ductus arteriosus, as determined by the investigator
4. Major congenital anomaly (e.g. congenital diaphragmatic hernia, congenital pulmonary adenomatoid malformation)
5. Meconium aspiration syndrome
6. Known allergy to any diuretic
7. Serum creatinine >1.7 mg/dL < 24 hours prior to first study dose
8. BUN >50 mg/dL < 24 hours prior to first study dose
9. Na <125 mmol/L < 24 hours prior to first study dose
10. K ≤2.5 mmol/L < 24 hours prior to first study dose
11. Ca ≤ 6 mg/dL < 24 hours prior to first study dose
12. Indirect bilirubin >10 mg/dL < 24 hours prior to first study dose
13. Any condition which would make the participant, in the opinion of the investigator, unsuitable for the study

Ages: 7 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2015-11-27 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Laughon, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill; Jason E Lang, MD, MPH, Study Chair — Duke University
Locations (21):
- United States (21):
  - Arkansas Children's Hospital/University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - University of Florida Jacskonville Shands Medical Center, Jacksonville, Florida
  - Wolfson Children's Hospital, Jacksonville, Florida
  - South Miami Hospital, South Miami, Florida
  - John's Hopkins Al Children's Hospital, St. Petersburg, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - Wesley Medical Center, Wichita, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Floating Hospital for Children at Tufts Medical Center, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Children's Mercy Hospital and Clinics, Kansas City, Missouri
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - The University of North Carolina at Chapel Hill/North Carolina Children's Hospital, Chapel Hill, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital/The Ohio State University, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Virginia Commonwealth University, Richmond, Virginia
  - West Virginia University, Morgantown, West Virginia

REFERENCES:
- [Derived] Greenberg RG, Lang J, Smith PB, Shekhawat P, Courtney SE, Hudak ML, Moya F, Iyengar A, Eldemerdash A, Bloom B, Go M, Hanna M, Rhein L, Aliaga S, Lewis T, Febre A, Kiefer AS, Bhatt-Mehta V, Khoury JA, Selewski D, Anand R, Martz K, Payne EH, Zimmerman KO, Benjamin DK Jr, Laughon M; Best Pharmaceuticals for Children Act - Pediatric Trials Network Steering Committee. Furosemide Safety in Preterm Infants at Risk for Bronchopulmonary Dysplasia: A Randomized Clinical Trial. J Pediatr. 2025 Aug;283:114629. doi: 10.1016/j.jpeds.2025.114629. Epub 2025 Apr 28. PMID 40306549

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Based on Cohort 2 safety data analysis, enrollment was stopped prior to Cohort 3.
Period: Overall Study
Arm/Group | Furosemide Cohort 1 | Placebo Cohort 1 | Furosemide Cohort 2 | Placebo Cohort 2 | Furosemide Cohort 3 | Placebo Cohort 3
Started | 32 | 10 | 30 | 10 | 0 | 0
Randomized, Not Dosed | 31 | 9 | 30 | 10 | 0 | 0
Pharmacokinetic (PK) Population | 20 | 0 | 19 | 0 | 0 | 0
Completed | 29 | 8 | 25 | 9 | 0 | 0
Not Completed | 3 | 2 | 5 | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 0 | 0 | 0
Not completed — Reason undisclosed | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Did not receive intervention | 1 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Based on Cohort 2 safety data analysis, enrollment was stopped prior to Cohort 3.
  Two participants in Cohort 1 were randomized, not dosed
Groups:
- Total: Total of all reporting groups
Arm/Group | Furosemide Cohort 1 | Placebo Cohort 1 | Furosemide Cohort 2 | Placebo Cohort 2 | Furosemide Cohort 3 | Placebo Cohort 3 | Total
Number analyzed (Participants) | 31 | 9 | 30 | 10 | 0 | 0 | 80
Age, Customized [Mean (Standard Deviation); unit: weeks]
  Gestational Age | 26.4 (1.4) | 26.3 (1.9) | 25.6 (1.4) | 25.5 (1.8) |  |  | 26.0 (1.5)
Age, Customized [Mean (Standard Deviation); unit: Days]
  Post Natal Age | 17 (7) | 18 (7) | 22 (6) | 24 (4) |  |  | 20 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 5 | 16 | 3 | 0 | 0 | 41
  Male | 14 | 4 | 14 | 7 | 0 | 0 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 7 | 2 | 0 | 0 | 12
  Not Hispanic or Latino | 28 | 8 | 22 | 8 | 0 | 0 | 66
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 7 | 9 | 3 | 0 | 0 | 29
  White | 18 | 2 | 16 | 6 | 0 | 0 | 42
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 3 | 0 | 4 | 0 | 0 | 0 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 9 | 30 | 10 | 0 | 0 | 80

OUTCOME MEASURES:

1. Primary Outcome: Safety as Determined by Adverse Events
Description: Safety was assessed following the initial study-specific procedure (e.g., screening blood draws, dosing) through 7 days post last study dose by frequency and incidence of adverse events and serious adverse events.
Time Frame: 35 days for each participant
Population: Based on Cohort 2 safety data analysis, enrollment was stopped prior to Cohort 3. Data are reported for the safety population.
Measure: Number; unit: Events
Groups:
- Furosemide Cohort 1: Within cohort 1, infants were randomized using a 3:1 scheme to receive furosemide or placebo. Those randomized to receive furosemide will receive 1mg/kg daily intravenously or 2 mg/kg daily enterally for 28 days.
  Furosemide Cohort 1: furosemide 1 mg/kg q 24 hours IV or 2 mg/kg q 24 hours enterally Cohorts will be enrolled sequentially after a safety review.
- Total: Sum of all groups
Arm/Group | Furosemide Cohort 1 | Placebo Cohort 1 | Furosemide Cohort 2 | Placebo Cohort 2 | Furosemide Cohort 3 | Placebo Cohort 3 | Total
Number analyzed (Participants) | 31 | 9 | 30 | 10 | 0 | 0 | 80
Events | 123 | 29 | 100 | 49 |  |  | 293

2. Secondary Outcome: Moderate-Severe BPD or Death Risk Throughout Weekly Treatment
Description: Moderate-severe BPD or death risk was defined by the NICHD Neonatal Research Network (NRN) BPD outcome estimator which provides an estimate of the risk of BPD (none, mild, moderate, severe) or death by postnatal day and is presented as a percentage. For this protocol, the categories were dichotomized to none-mild vs. moderate-severe-death. The risk of BPD or death was defined by the NICHD NRN BPD estimator on days 7, 14, 21 and 28 of study drug using the closest day available from the BPD estimator. The BPD estimator includes infants up to 28 postnatal days; for infants in this protocol older than that, 28-day estimates are used.
Time Frame: Risk measured weekly through Week 4
Population: Data are reported for the safety population. Overall 82 participants were randomized, but 2 were not dosed. 80 participants were analyzed for BPD status.
  Based on Cohort 2 safety data analysis, enrollment was stopped prior to Cohort 3.
Measure: Mean (Standard Deviation); unit: percent probability of BPD or death risk
Groups:
- Weekly Total: Weekly total (Cohort 1 Furosemide/Placebo and Cohort 2 Furosemide/Placebo
Arm/Group | Furosemide Cohort 1 | Placebo Cohort 1 | Furosemide Cohort 2 | Placebo Cohort 2 | Furosemide Cohort 3 | Placebo Cohort 3 | Weekly Total
Number analyzed (Participants) | 31 | 9 | 30 | 10 | 0 | 0 | 80
percent probability of BPD or death risk
  Week 0: number analyzed (Participants) | 29 | 9 | 29 | 10 | 0 | 0 | 77
  Week 0 | 57.9 (20.5) | 52.8 (23.0) | 66.7 (16.8) | 70.9 (22.2) |  |  | 62.3 (20.2)
  Week 1: number analyzed (Participants) | 29 | 9 | 27 | 10 | 0 | 0 | 75
  Week 1 | 55.4 (21.2) | 55.5 (20.6) | 65.9 (17.5) | 71.6 (20.4) |  |  | 61.4 (20.3)
  Week 2: number analyzed (Participants) | 27 | 9 | 25 | 10 | 0 | 0 | 71
  Week 2 | 52.1 (23.3) | 56.2 (21.8) | 61 (18.3) | 65.0 (18.4) |  |  | 57.6 (20.9)
  Week 3: number analyzed (Participants) | 26 | 8 | 24 | 10 | 0 | 0 | 68
  Week 3 | 52.1 (28) | 40.4 (25.2) | 61.3 (18.2) | 57.9 (30.7) |  |  | 54.9 (25.4)
  Week 4: number analyzed (Participants) | 23 | 8 | 20 | 9 | 0 | 0 | 60
  Week 4 | 44.0 (23.6) | 40.9 (27.9) | 53.0 (20.6) | 54.4 (34.1) |  |  | 48.2 (25.0)

3. Secondary Outcome: Number of Participants With Moderate-Severe BPD or Death Risk as Clinically Determined
Description: Moderate-severe BPD or death risk was defined using the NICHD Neonatal Research Network BPD outcome estimator.
Time Frame: 36 weeks postmenstrual age
Population: Data are reported for the safety population. Based on Cohort 2 safety data analysis, enrollment was stopped prior to Cohort 3.
Measure: Count of Participants; unit: Participants
Arm/Group | Furosemide Cohort 1 | Furosemide Cohort 2 | Placebo Cohort 1 | Placebo Cohort 2 | Furosemide Cohort 3 | Placebo Cohort 3
Number analyzed (Participants) | 31 | 30 | 9 | 10 | 0 | 0
Participants | 17 | 22 | 6 | 6 |  |

4. Secondary Outcome: Clearance
Description: Data was collected from Furosemide/Active Cohort 1 and Cohort 2 and combined Cohorts. In total 39 active drug recipients participated. PK samples were collected after 7 days on study drug at recommended time points through 28 days on study drug plus one elimination (post drug discontinuation) time point.
Time Frame: After study drug administration completion within 30 minutes, 2-4 hours, 6-8 hours, 12-16 hours, and 20-22 hours; within 30 minutes prior to the next dose; and within 48-72 hours of the final study drug administration.
Population: Data was collected from the Furosemide cohort 1 and 2, and combined. In total 39 active drug recipients participated in the population PK.
Measure: Median (Full Range); unit: (mL/h/kg)
Groups:
- Furosemide Cohort 1: PK Population: Furosemide/Active drug arms from Cohort 1
- Furosemide Cohort 2: PK Population: Furosemide/Active drug arms from Cohort 2
- Furosemide (Cohort 1 and Cohort 2): PK Population: Furosemide/Active drug arms from Cohort 1 and Cohort 2
Arm/Group | Furosemide Cohort 1 | Furosemide Cohort 2 | Furosemide (Cohort 1 and Cohort 2)
Number analyzed (Participants) | 20 | 19 | 39
(mL/h/kg) | 16.3 [3.7 to 36] | 21.8 [7.7 to 43.6] | 18 [3.7 to 43.6]

5. Secondary Outcome: Volume of Distribution
Description: as for outcome 4
Time Frame: as for outcome 4
Population: Data was collected from the Furosemide Cohort 1 and Cohort 2 and combined. In total, 39 active drug recipients participated in the population PK.
Measure: Median (Full Range); unit: mL
Groups:
- Furosemide All (Cohort 1 and Cohort 2): PK Population: Furosemide/Active drug arms from Cohort 1 and Cohort 2
Arm/Group | Furosemide Cohort 1 | Furosemide Cohort 2 | Furosemide All (Cohort 1 and Cohort 2)
Number analyzed (Participants) | 20 | 19 | 39
mL | 236.7 [148.9 to 366.5] | 242.8 [148.9 to 380.2] | 242.8 [149.2 to 380.2]

6. Secondary Outcome: Half-life
Description: as for outcome 4
Time Frame: as for outcome 4
Population: Data were collected from the two Furosemide cohorts and the combined analysis includes all 39 active drug recipients who participated in the population PK .
Measure: Median (Full Range); unit: hours
Groups:
- Furosemide Cohort 1: PK Population: Furosemide/Active drug from Cohort 1
- Furosemide Cohort 2: PK Population: Furosemide/Active drug from Cohort 2
- Furosemide Cohort 1 and Cohort 2: PK Population: Combined Furosemide/Active drug from Cohort 1 and Cohort 2
Arm/Group | Furosemide Cohort 1 | Furosemide Cohort 2 | Furosemide Cohort 1 and Cohort 2
Number analyzed (Participants) | 20 | 19 | 39
hours | 9.8 [4.4 to 43.5] | 7.3 [3.6 to 20.6] | 8.8 [3.6 to 43.5]

7. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve
Description: Population PK data were collected from the two Furosemide cohorts and includes all 39 active drug recipients.
Time Frame: as for outcome 4
Population: Data was collected from Furosemide/Active Cohort 1 and Cohort 2 and combined Cohorts. In total 39 active drug recipients participated. PK samples were collected after 7 days on study drug at recommended time points through 28 days on study drug plus one elimination (post drug discontinuation) time point.
Measure: Median (Full Range); unit: mg*h/L
Groups:
- Furosemide (Cohort 1 and Cohort 2): PK Population: Furosemide/Active drug from Cohort 1 and Cohort 2
Arm/Group | Furosemide Cohort 1 | Furosemide Cohort 2 | Furosemide (Cohort 1 and Cohort 2)
Number analyzed (Participants) | 20 | 19 | 39
mg*h/L | 2165 [1011 to 6059] | 6016 [2801 to 12330] | 4639 [1011 to 12330]

ADVERSE EVENTS:
Time Frame: Following provision of Informed consent through final assessment, a total of approximately 35 days.
Description: Based on Cohort 2 safety data analysis, enrollment was stopped prior to Cohort 3.
Arm/Group | Furosemide Cohort 1 | Placebo Cohort 1 | Furosemide Cohort 2 | Placebo Cohort 2 | Furosemide Cohort 3 | Placebo Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/9 | 1/30 | 0/10 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 5/31 | 1/9 | 6/30 | 0/10 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 28/31 | 9/9 | 28/30 | 9/10 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Furosemide Cohort 1 (N=31) | Placebo Cohort 1 (N=9) | Furosemide Cohort 2 (N=30) | Placebo Cohort 2 (N=10) | Furosemide Cohort 3 (N=0) | Placebo Cohort 3 (N=0)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | NA | NA | NA
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Meningitis herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Necrotising colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | NA | NA | NA
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | NA | NA | NA
Necrotising colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Respiratory failure (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Respiratory track infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA | NA
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Furosemide Cohort 1 (N=31) | Placebo Cohort 1 (N=9) | Furosemide Cohort 2 (N=30) | Placebo Cohort 2 (N=10) | Furosemide Cohort 3 (N=0) | Placebo Cohort 3 (N=0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0
Chronic Respiratory Disease (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 0 (0) | 1 (1) | 1 (1) | NA | NA
Anaemia neonatal (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | NA | NA
Bandaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | NA | NA
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 3 (3) | 0 (0) | 4 (5) | 1 (1) | NA | NA
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Retinopathy of prematurity (Eye disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | NA | NA
abdominal distension (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | NA | NA
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | NA | NA
Necrotising colitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | NA | NA
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | NA | NA
Pneumonia escherichia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | NA | NA
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | NA | NA
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | NA | NA
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Blood bicarbonate increased (Investigations) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | NA | NA
Blood creatinine increased (Investigations) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | NA | NA
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | NA | NA
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | NA | NA
Bilirubin conjugate increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Blood sodium decreased (Investigations) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | NA | NA
Blood urea increased (Investigations) | 0 (0) | 8 (8) | 0 (0) | 0 (0) | NA | NA
Cardiac murmur (Investigations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Chest X-ray abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Sputum culture positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Electrolyte imbalance (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | NA | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | NA | NA
Hyperphosphataemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 4 (5) | 1 (1) | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 10 (10) | 1 (1) | 7 (8) | 0 (0) | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | NA | NA
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | NA | NA
Growth retardation (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | NA | NA
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Hypertonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Periventricular leukomalacia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Seizure (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | NA | NA
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | NA | NA
Testicular swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | NA | NA
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | NA | NA
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | NA | NA
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | NA | NA
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | NA | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | NA | NA
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-09-27): https://cdn.clinicaltrials.gov/large-docs/98/NCT02527798/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT02527798/SAP_001.pdf